CLINICAL TRIAL: NCT05025020
Title: Incorporating Three-Dimensional Visualization in Breast Reconstruction Consultation
Brief Title: Use of an Interactive 3D Tool During Consultation for Breast Reconstruction Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-318
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Reconstruction Surgery; Interactive 3D Tool; Consultation; 21-318
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard consultation with interactive 3D visualization (Experimental): Participants in this group will use the interactive 3D tool in addition to receiving the standard surgical consultation before their breast reconstruction procedure.
  Interventions: Other: interactive 3D tool; Other: BREAST-Q Reconstruction Module; Other: DQI; Other: Ottawa Decision Regret Scale
- Standard consultation (Active Comparator): Participants in this group will receive a standard surgical consultation before their breast reconstruction procedure.
  Interventions: Other: BREAST-Q Reconstruction Module; Other: DQI; Other: Ottawa Decision Regret Scale

INTERVENTIONS:
Other: interactive 3D tool — The study tool displays 3-dimensional step-by-step animations of autologous and implant-based breast reconstruction procedures.
  Arms: Standard consultation with interactive 3D visualization
Other: BREAST-Q Reconstruction Module — The BREAST-Q Reconstruction Module1-3 has 6 domains that cover various aspects of patient satisfaction and quality of life. BREAST-Q is part of our standard of care for patients treated for breast cancer and referred for reconstruction.
Other: DQI — The DQI has 3 domains that cover decision-specific questions about what it is like for a patient to make decisions about reconstruction after breast cancer treatment.
Other: Ottawa Decision Regret Scale — The validated Decision Regret Scale measures distress or remorse after a health care decision by the use of 5 items to indicate the extent to which the respondent agrees or disagrees with the statements in the regret scale.

SUMMARY:
The purpose of this study is to find out whether using an interactive 3D tool during a standard surgical consultation can lead to greater patient satisfaction with the information provided about breast reconstruction options than the standard consultation alone. The study researchers will also assess whether women whose surgical consultation includes the use of the 3D tool are more satisfied with their breasts and with the decisions they made about their reconstruction procedure.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Presenting at MSK for initial breast reconstruction consultation
* Planning to undergo mastectomy at time of consultation
* English spoken as primary language
* Able to provide informed consent without a legally authorized representative

Exclusion Criteria:

* Prior breast reconstruction
* Prior breast reconstruction consultation with a plastic surgeon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 88 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
BREAST-Q Satisfaction | 4 weeks
  scores at 4 weeks (T2) Scores for each domain of the BREAST-Q range from 0 to 100, implying a continuum of increasing satisfaction or better quality of life.

SECONDARY OUTCOMES:
BREAST-Q Satisfaction | 3 months after surgery
  The outcome will be the score (continuous variable ranging from 0 to 100 for linear regression or ordinal categories, ranging from 1 to 4 for ordinallogistic regression, where 1 represents lowest satisfaction and 4 represents highest satisfaction), and the primary predictor of interest will be type of consultation provided.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Stern, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
URL: http://www.mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm